CLINICAL TRIAL: NCT05648630
Title: Improving Exercise Rehabilitation Efficacy and Outcomes in Veterans With Peripheral Artery Disease: Targeting Oxidative Stress and Inflammation
Brief Title: Improving Exercise Rehabilitation Efficacy Outcomes Veterans Peripheral Artery Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate participant recruitment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E3913-W; RX003913 (Other Grant/Funding Number: Department of Veterans Affairs ORD)
Record Dates: First submitted 2022-11-04; First posted 2022-12-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Artery Disease (D058729); Oxidative Stress (D018384); Inflammation (D007249)
Keywords: inflammation (D007249); Skeletal muscle (D018482); Antioxidants (D000975)
MeSH Terms: conditions — Peripheral Arterial Disease; Inflammation | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Two separate groups of subjects (patients with PAD) receiving PB125 or Placebo
Masking Description: Two separate groups of subjects (patients with PAD) receiving PB125 or Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Rehabilitation+PB125 (Experimental): Participants will be assigned to the Exercise+Placebo or Exercise+PB125 rehabilitation interventions using block randomization.
  Interventions: Dietary Supplement: PB125; Behavioral: Exercise Rehabilitation
- Exercise Rehabilitation with Placebo (Placebo Comparator): Participants will be assigned to the Exercise+Placebo rehabilitation interventions using block randomization.
  Interventions: Dietary Supplement: Placebo; Behavioral: Exercise Rehabilitation

INTERVENTIONS:
Dietary Supplement: PB125 — PB125 is a naturally-derived plant-based supplement that activates the Nuclear Factor Erythroid-2-like 2 (Nrf2) system to stimulate induction of endogenous antioxidants and anti-inflammatory pathways.
  Arms: Exercise Rehabilitation+PB125
Dietary Supplement: Placebo — A placebo will be used in combination with exercise rehabilitation allowing for a double blinded placebo controlled design.
  Arms: Exercise Rehabilitation with Placebo
Behavioral: Exercise Rehabilitation — A 12-week treadmill based supervised rehabilitation

SUMMARY:
Physical activity is the most beneficial and cost-effective treatment for Veterans with PAD, however, issues with oxygen delivery and utilization dramatically impair exercise compliance. The cause of these oxygen delivery and utilization impairments is likely increased oxidative stress and inflammation. The proposed project will comprehensively examine the novel strategy of Nuclear Factor Erythroid-2-like 2 (Nrf2) activation using PB125, aimed at diminishing oxidative stress and inflammation, and thereby lessening the negative impacts of the disease. This therapeutic will be evaluated in isolation and in combination with exercise rehabilitation to determine if there is a complimentary benefit. The ultimate goal is to provide insight into a potential novel therapeutic treatment for this disease, therefore, improving exercise tolerance and quality of life in this growing population.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a debilitating atherosclerotic disease caused by plaque development in the arteries leading to diminished skeletal muscle blood flow, oxygen delivery, and metabolic dysfunction during ambulation causing marked exercise intolerance. Veterans have a disproportionate risk of developing PAD compared to the general population because of higher levels of smoking, hypertension, diabetes, and obesity. Worryingly, the mortality rate for PAD in Veterans (~30%) is nearly double that of the general population. Currently, the best treatment of PAD is exercise rehabilitation, however, issues with patient motivation and pain reduce the effectiveness of this treatment. There is a pressing, and unmet need to identify the sites and underlying mechanisms of the systemic dysfunction leading to exercise intolerance induced by PAD. Oxidative stress and inflammation play important roles in the development and progression of PAD. Critically, the peripheral vasculature (diminished blood flow) and mitochondria (diminished respiration) are primary determinants/mechanisms responsible for exercise intolerance in health and disease that are particularly vulnerable to elevations in oxidative stress and inflammation, making these likely sites of systemic dysfunction leading to exercise intolerance in Veterans with PAD. Any vascular or mitochondrial dysfunction would further augment oxidative stress and inflammation initiating a vicious cycle. It is the central hypothesis that increased endogenous antioxidant capacity and diminished inflammation will improve oxygen delivery and utilization during exercise, thus, increasing the efficacy of exercise rehabilitation due to increased adherence and exercise capacity. To test this hypothesis, the investigators will utilize the naturally-derived Nuclear Factor Erythroid-2-like 2 (Nrf2; the "master regulator of antioxidant enzymes") activator, PB125, to stimulate induction of endogenous antioxidants and decrease the activity of inflammatory pathways. Veterans with PAD will be randomly assigned to receive either PB125 or Placebo supplementation. Each Veteran will undergo three phases of testing: 1) baseline, 2) post 1 month of supplement loading, and 3) post 12 weeks of exercise rehabilitation with continued supplementation. Functional capacity and cognitive function (Aim 1), Vascular function and exercising hemodynamics (Aim 2), and in vivo and ex vivo mitochondrial respiration (Aim 3) will be assessed each phase. Monthly assessments of functional capacity, behavioral regulation, quality of life, and physical activity will track improvements across the trial. At the conclusion of these studies, the investigators will have expanded the knowledge of the mechanisms underlying exercise intolerance in Veterans suffering from PAD, and, more importantly from a clinical perspective, provided insight into a potential novel therapeutic treatment to improve exercise rehabilitation efficacy for this population. It is anticipated this advancement will contribute to advancing clinical practice in rehabilitative medicine, and ultimately, improving the quality of life for Veterans living with PAD.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 and older with clinically diagnosed femoropopliteal PAD (ankle-brachial index < 0.9)
* Must understand the study requirements and be willing and able to sign an informed consent document
* Patients with mild cognitive impairment (i.e., montreal cognitive assessment (MOCA) <26) will be included but must have a responsible caregiver or spouse present during the informed consent
* Women that are not pregnant, breastfeeding, or likely to become pregnant within the next 6 months

Exclusion Criteria:

* Patients with a bleeding disorder that would contraindicate the performance of a muscle biopsy, such as a history of clinically significant bleeding diathesis (i.e., Hemophilia A or B, Von Willebrand's Disease, or congenital Factor VII deficiency)
* Patients with a complex atherosclerotic lesion such that withholding medication creates disproportionate risk
* Women currently taking hormone replacement therapy
* Any other condition or event considered exclusionary by the PI and faculty physician

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Six-minute Walk Test (6MWT) Change | Baseline, month 1, month 2, month 3, month 4
  6MWT will be quantified with total distance, last minute speed, and claudication onset time. Greater distance and higher speed indicates better functional capacity and greater change over time suggests improvement.
Exercise pressor response (EPR) Change | Baseline, month 1, month 2, month 3, month 4
  EPR will be quantified with the change in mean arterial blood pressure from rest to exercise. A greater EPR indicates elevated cardiovascular risk and a reduction in the EPR over time suggests improvement.
Intramuscular maximal bioenergetics (Vmax) Change | Baseline, month 1, month 4
  Vmax will be quantified as the rate of intramuscular phosphocreatine replenishment following exercise. A greater Vmax indicates better mitochondrial and hemodynamic function and greater change over time suggests improvement.

CONTACTS AND LOCATIONS:
Overall Officials: David W. Wray, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (2):
- United States (2):
  - University of Utah Dept of Vascular Surgery, Salt Lake City, Utah
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Upon written request, a limited, de-identified, anonymized dataset will be created pursuant to the Data Use Agreement. This DUA will limit the use of the dataset and prohibit the recipient from taking steps to identify individuals whose data is included in the dataset. This dataset will be provided through a password-protected, machine-readable database format. Whenever possible, the dataset will be delivered through physical transfer of the storage medium.